CLINICAL TRIAL: NCT02890108
Title: Effect of Consumption of Non Caloric Sweeteners and Insulin Sensibility
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Instituto de Nutrición y Tecnología de los Alimentos (Other)
Responsible Party: Principal Investigator, Romina Goza Ferreira, magister thesis student in adult clinical nutrition, Instituto de Nutrición y Tecnología de los Alimentos
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: EANC-1
Record Dates: First submitted 2016-08-19; First posted 2016-09-07 (Estimated); Last update posted 2016-09-07 (Estimated); Status verified 2016-08

CONDITIONS: Insulin Sensitivity
Keywords: High-Intensity Sweeteners; Non-Nutritive Sweeteners; Artificial sweeteners; Glucose intolerance
MeSH Terms: conditions — Insulin Resistance; Glucose Intolerance | interventions — Sugar-Sweetened Beverages; Artificially Sweetened Beverages

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Sugar sweetened beverages (Experimental): Subjects will receive, in 3 different ocassions, 350cc (1 can) of a sugar sweetened beverage, that contain 38,7 grams of carbs and 154 kcal, separated by at least 1 week each one
  Interventions: Dietary Supplement: Sugar sweetened beverages
- Artificially sweetened beverage (Experimental): Subjects will receive, in 3 different ocassions, 350cc (1 can) of a artificially sweetened beverage, that contain 84 mg of Aspartame, 56 mg of Acesulfame K and 0,7 kcal, separated by at least 1 week each one
  Interventions: Dietary Supplement: Artificially sweetened beverages

INTERVENTIONS:
Dietary Supplement: Sugar sweetened beverages — 350 cc (1 can) of sugar sweetened beverage
  Other Names: Sugar sweetened drinks
  Arms: Sugar sweetened beverages
Dietary Supplement: Artificially sweetened beverages — 350 cc (1 can) of artificially sweetened beverage
  Other Names: Artificially sweetened drinks
  Arms: Artificially sweetened beverage

SUMMARY:
This study will compare the effect of acute consumption of two carbonated drinks, sweetened with sugar or with non-caloric sweeteners, over the insulin response of healthy adults who normally consumed foods or drinks that contain non-caloric sweeteners

DETAILED DESCRIPTION:
During the last decades there has been a sustained increase in prevalence of overweight and obesity and, along with it, of chronic noncommunicable diseases. There have been addressed various management strategies, including sugar replacement for Non-caloric Artificial Sweeteners (NAS). Nevertheless, in several cohort studies it has found the opposite effect, it has observed associations between the consumption of NAS with greater weight gain and increased risk of type 2 diabetes and metabolic syndrome. In clinical trials, in both humans and mice, there has been greater association with glucose intolerance, being 3 possible mechanisms: 1) dysbiosis of the intestinal microbiota; 2) altered regulation of appetite cephalic phase and secretion of glucagon like peptide-1 (GLP-1); and 3) increased intestinal glucose absorption via increased Sodium-Glucose Linked Transporter-1 (SGLT-1) and Glucose transporter 2 (GLUT2), transporters to glucose absorption.

In the following review the major findings in the literature regarding the consumption of NAS and its deleterious effects on human health will be studied.

ELIGIBILITY:
Inclusion Criteria:

* Body Mass Index (BMI) between 18,5 - 24,9 kg/mt2
* Healthy men or women
* Fasting plasma glucose < 100 mg/dL

Exclusion Criteria:

* Consumption of drugs affecting glucose metabolism, antihypertensives or lipid lowering
* Subjects with insulin resistance, type 1 or 2 diabetes, dyslipidemia, hypertension; heart, liver or kidney disease, respiratory failure, stroke, or any chronic illness.
* Pregnant women.
* Being treated to gain or lose weight.
* History of recurrent episodes of acute diarrhea.

Ages: 25 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Estimated)
Dates: Start 2016-08; Primary Completion 2016-09 (Estimated); Study Completion 2016-10 (Estimated)

PRIMARY OUTCOMES:
Insulin sensibility | Measured at 6 intervals (3 times sugar sweetened beverages and 3 times artificially sweetened beverages), separated at least by 1 week from each other. All the tests must be assessed during 10 weeks utmost.
  One insulinemic curve will be conducted to assess the effect of consumption of artificially sweetened beverage on insulin response compared to the consumption of a sugar sweetened drink.

SECONDARY OUTCOMES:
Glycemic response | Measured at 6 intervals (3 times sugar sweetened beverages and 3 times artificially sweetened beverages), separated at least by 1 week from each other. All the tests must be assessed during 10 weeks utmost.
  One glycemic curve will be conducted to assess the effect of consumption of artificially sweetened beverage on glycemic response compared to the consumption of a sugar sweetened drink.

CONTACTS AND LOCATIONS:
Overall Officials: Romina A Goza Ferreira, Magister c, Principal Investigator — Institute of Nutrition and Tecnology of Food, University of Chile; Sandra Hirsch Birn, Magister, Study Director — Institute of Nutrition and Tecnology of Food, University of Chile
Locations (1):
- Institute of Nutrition and Tecnology of Food, University of Chile, Santiago, Metropolitan Region, Chile

IPD SHARING:
Plan to Share IPD: No
All the data is confidential and only will be show if ethics committee ask for it

REFERENCES:
- [Background] Pan A, Malik VS, Hao T, Willett WC, Mozaffarian D, Hu FB. Changes in water and beverage intake and long-term weight changes: results from three prospective cohort studies. Int J Obes (Lond). 2013 Oct;37(10):1378-85. doi: 10.1038/ijo.2012.225. Epub 2013 Jan 15. PMID 23318721
- [Background] de Koning L, Malik VS, Rimm EB, Willett WC, Hu FB. Sugar-sweetened and artificially sweetened beverage consumption and risk of type 2 diabetes in men. Am J Clin Nutr. 2011 Jun;93(6):1321-7. doi: 10.3945/ajcn.110.007922. Epub 2011 Mar 23. PMID 21430119
- [Background] Nettleton JA, Lutsey PL, Wang Y, Lima JA, Michos ED, Jacobs DR Jr. Diet soda intake and risk of incident metabolic syndrome and type 2 diabetes in the Multi-Ethnic Study of Atherosclerosis (MESA). Diabetes Care. 2009 Apr;32(4):688-94. doi: 10.2337/dc08-1799. Epub 2009 Jan 16. PMID 19151203
- [Background] Pepino MY. Metabolic effects of non-nutritive sweeteners. Physiol Behav. 2015 Dec 1;152(Pt B):450-5. doi: 10.1016/j.physbeh.2015.06.024. Epub 2015 Jun 19. PMID 26095119
- [Background] Swithers SE. Artificial sweeteners produce the counterintuitive effect of inducing metabolic derangements. Trends Endocrinol Metab. 2013 Sep;24(9):431-41. doi: 10.1016/j.tem.2013.05.005. Epub 2013 Jul 10. PMID 23850261
- [Background] Feijo FM, Ballard CR, Foletto KC, Batista BAM, Neves AM, Ribeiro MFM, Bertoluci MC. Saccharin and aspartame, compared with sucrose, induce greater weight gain in adult Wistar rats, at similar total caloric intake levels. Appetite. 2013 Jan;60(1):203-207. doi: 10.1016/j.appet.2012.10.009. Epub 2012 Oct 23. PMID 23088901
- [Background] Anton SD, Martin CK, Han H, Coulon S, Cefalu WT, Geiselman P, Williamson DA. Effects of stevia, aspartame, and sucrose on food intake, satiety, and postprandial glucose and insulin levels. Appetite. 2010 Aug;55(1):37-43. doi: 10.1016/j.appet.2010.03.009. Epub 2010 Mar 18. PMID 20303371
- [Background] Suez J, Korem T, Zeevi D, Zilberman-Schapira G, Thaiss CA, Maza O, Israeli D, Zmora N, Gilad S, Weinberger A, Kuperman Y, Harmelin A, Kolodkin-Gal I, Shapiro H, Halpern Z, Segal E, Elinav E. Artificial sweeteners induce glucose intolerance by altering the gut microbiota. Nature. 2014 Oct 9;514(7521):181-6. doi: 10.1038/nature13793. Epub 2014 Sep 17. PMID 25231862
- [Background] Palmnas MS, Cowan TE, Bomhof MR, Su J, Reimer RA, Vogel HJ, Hittel DS, Shearer J. Low-dose aspartame consumption differentially affects gut microbiota-host metabolic interactions in the diet-induced obese rat. PLoS One. 2014 Oct 14;9(10):e109841. doi: 10.1371/journal.pone.0109841. eCollection 2014. PMID 25313461
- [Background] Brown RJ, Walter M, Rother KI. Ingestion of diet soda before a glucose load augments glucagon-like peptide-1 secretion. Diabetes Care. 2009 Dec;32(12):2184-6. doi: 10.2337/dc09-1185. Epub 2009 Oct 6. PMID 19808921
- [Background] Temizkan S, Deyneli O, Yasar M, Arpa M, Gunes M, Yazici D, Sirikci O, Haklar G, Imeryuz N, Yavuz DG. Sucralose enhances GLP-1 release and lowers blood glucose in the presence of carbohydrate in healthy subjects but not in patients with type 2 diabetes. Eur J Clin Nutr. 2015 Feb;69(2):162-6. doi: 10.1038/ejcn.2014.208. Epub 2014 Oct 1. PMID 25271009
- [Background] Pepino MY, Tiemann CD, Patterson BW, Wice BM, Klein S. Sucralose affects glycemic and hormonal responses to an oral glucose load. Diabetes Care. 2013 Sep;36(9):2530-5. doi: 10.2337/dc12-2221. Epub 2013 Apr 30. PMID 23633524